CLINICAL TRIAL: NCT07015476
Title: Retrospective Observational Evaluation of the Bone Mineral Density Outcome of Different Oestrogen Therapy Regimens in Young Women With Amenorrhea
Brief Title: Retrospective Observational Evaluation of the Bone Mineral Density Outcome in Young Women With Amenorrhea
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: AMEN-20
Record Dates: First submitted 2024-12-30; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-11

CONDITIONS: Amenorrhea
Keywords: Amenorrhea; Bone Mass; Estrogen Therapy
MeSH Terms: conditions — Amenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GROUP A: Natural estrogen (estradiol or valerate estradiol) administered transdermically
- GROUP B: Natural estrogen administered orally
- GROUP C: Etinil-estradiol administered orally
- GROUP D: No therapy

SUMMARY:
The study aims to evaluate the outcomes of different estrogen therapy regimens in patients with amenorrhea who face prolonged periods of hypoestrogenism.

The primary objective is to compare the outcomes on bone mass of different therapeutic regimens and identify more favorable. For this purpose, densitometry parameters such as BMD, T-score and Z-score at the level of the lumbar spine, femur and entire skeleton will be considered, comparing a bone densitometry (DXA technique, Dual X-ray Absorptiometry) Baseline with one carried out after at least one year of therapy. The secondary objective of the study is to assess other systemic/metabolic implications of the different therapies.

DETAILED DESCRIPTION:
The present retrospective monocentric observational study involves the recruitment of patients afferite at the U.O. of Gynecology and Physiopathology of Human Reproduction in the time interval between 2011 and 2020 in condition of amenorrhea greater than 6 months, Aged between 15 and 39 at the time of first visit.

Patients will be asked to participate in this study during the outpatient follow-up visit.

The study will involve data collection through consultation of health records.

The objectives of the study will therefore be achieved by analysing the following parameters, which can be fully deduced from the medical records of the subjects in the study:

* Collection of anamnestic (eating habits and sports, pathologies of note, taking drugs, previous surgical interventions, smoking habit, gynecological history).
* Physical examination: calculation of BMI, acne and hirsutism score (GAGS and Ferriman score), blood pressure measurement, gynecological physical examination
* Transvaginal or transabdominal pelvic ultrasound
* Lumbar, femoral, total body dual-energy x-ray absorptiometry (DXA)
* Blood tests (blood count, lipid profile, glycemic, liver, kidney, hormonal status)
* Reports of other visits and specialist examinations performed by the patients brought to view during the visit

ELIGIBILITY:
Inclusion criteria:

* Patients who have presented themselves to the O.U. of Gynecology and Human Reproduction Pathophysiology in the period from 2011 to 2020 with amenorrhea over 6 months, and aged between 15 and 39 years at the time of the visit.
* Patients who have reached the age of 18 at the time of surgery.
* Patients for whom informed consent has been obtained.

Exclusion criteria: No exclusion criteria are provided.

Ages: 15 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The present retrospective observational study, monocentric, involves the recruitment of patients who have presented themselves to the U.O. of Gynecology and Pathophysiology of Human Reproduction in the time interval between 2011 and 2020 in condition of amenorrhea above 6 months, Aged between 15 and 39 at the time of first visit. Patients will be asked to participate in this study during the outpatient follow-up visit.
  The study will involve data collection through consultation of health records.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Until the end of the study (1 year)
  The objectives of the study will be achieved by analysing the following parameters:
  Collection of anamnestic (eating habits and sports, pathologies of importance, medication intake, previous surgical interventions, smoking habit, gynecological history).
Primary Outcome Measure | Until the end of the study (1 year)
  The objectives of the study will be achieved by analysing the following parameters: Physical examination: calculation of BMI (weight Kg/(height meters * height in meters), blood pressure (mm Hg)
Primary Outcome Measure | Until the end of the study (1 year)
  The objectives of the study will be achieved by analysing the following parameters: Transvaginal or transabdominal pelvic ultrasound (Uterus measures mm; endometrium thickness mm; ovary size volume cc and mesures mm)
Primary Outcome Measure | Until the end of the study (1 year)
  The objectives of the study will be achieved by analysing the following parameters:
  Lumbar, femoral, total body dual-energy x-ray absorptiometry (DXA): BMD (g/cm2); T score e Z score.
Primary Outcome Measure | Until the end of the study (1 year)
  Blood tests: hemoglobin (g/gl), hematocrit (%),red blood cells (million/µl), Platelets (x1000/ µl), Glucose (mg/dl), Alt (U/L), Ast (U/L), triglycerides (mg/dl), Total cholesterol (mg/dl), HDL Cholesterol (mg/dl), LH (mU/ml), FSH (mU/ml), Testosteron (ng/ml), Proladctin ( ng/ml), Estradiol (pg/ml); Urinalysis: PH, proteins(mg/dl) Glucose (mg/dl), Red blood cells (num/microL), Leukocytes

SECONDARY OUTCOMES:
GAGs and Ferriman Score | Until the end of the study (1 year)
  For Acne: The GAGS divides the face (forehead, each cheek, nose, and chin), chest, and back into six areas, and the severity in each zone is then assessed on a scale of 0 to 4 (0, no lesions; 1, comedones; 2, papules; 3, pustules; and 4, nodules.
GAGs and Ferriman Score | Until the end of the study (1 year)
  For Hirsutism: The Ferriman-Gallwey is widely used to evaluate and quantify hirsutism in women. The method incorporates nine body regions (excludes legs and forearms) for the assessment of hair growth, rated from 0 (no growth of terminal hair) to 4 (extensive hair growth) in each of the nine locations.
  The total score therefore can range from 0 to 36 and a score of > 8 is considered a sign of androgen excess in Caucasian women. A score of 8 -15 indicates mild hirsutism and >15 indicates moderate or severe hirsutism. For other ethnic groups, the amount of hair expected for that ethnicity should be considered.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Meriggiola, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero -Univeristaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No